CLINICAL TRIAL: NCT03438539
Title: Brief Online Interventions for Alcohol Use: A Crowdsourced Study
Brief Title: Brief Online Interventions for Alcohol Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Rush (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Craig Rush, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mTurk 10; R34DA038869 (NIH)
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Results first posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: An Internet survey hosted by Amazon.com's Mechanical Turk and Qualtrics: Online Survey Software will be used in this protocol. Cognitive tasks will be coded using PsyToolKit, an open-source tool for programming and running cognitive-psychological experiments and surveys online (Stoet, 2017). A mixed-model design will be used such that subjects are randomly assigned to one of three cognitive training conditions and two information feedback conditions (i.e., between-subjects variables). The same subjects will be sampled at each time point in the study (i.e., repeated/longitudinal variables).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Attentional Control with Normative Feedback (Sham Comparator): Control training tasks will include completion of basic arithmetic problems for approximately 5 minutes. Subjects assigned to normative feedback will be directed to a statement standardized based on subjects' reported average number of standard drinks per week, age, and gender.
  Interventions: Behavioral: Normative Feedback
- Inhibitory Control Training with Normative Feedback (Experimental): The inhibitory control training task is a modified version of the Cued Go/No-Go tasks (Weafer and Fillmore, 2012; Miller et al. 1991) and is based on a task currently used in our laboratory targeting cocaine inhibitory control. Subjects assigned to normative feedback will be directed to a statement standardized based on subjects' reported average number of standard drinks per week, age, and gender.
  Interventions: Behavioral: Normative Feedback; Behavioral: Inhibitory Control Training
- Working Memory Training with Normative Feedback (Experimental): A battery of working memory tasks will be used during the intervention period. These tasks were selected from previous research evaluating working memory training in substance use disorder (Bickel et al., 2011b; Houben et al., 2011b). Tasks will include visuospatial working memory task, digit span task, letter span task, and the n-back task. Subjects assigned to normative feedback will be directed to a statement standardized based on subjects' reported average number of standard drinks per week, age, and gender.
  Interventions: Behavioral: Normative Feedback; Behavioral: Working Memory Training
- Attentional Control without Normative Feedback (No Intervention): Control training tasks will include completion of basic arithmetic problems for approximately 5 minutes. Subjects assigned to not receive normative feedback will receive feedback on time spent doing a non-alcohol related activity as an attention/informational control (e.g., time spent watching television; LaBrie et al., 2013).
- Inhibitory Control Training without Normative Feedback (Experimental): The inhibitory control training task is a modified version of the Cued Go/No-Go tasks (Weafer and Fillmore, 2012; Miller et al. 1991) and is based on a task currently used in our laboratory targeting cocaine inhibitory control. Subjects assigned to not receive normative feedback will receive feedback on time spent doing a non-alcohol related activity as an attention/informational control (e.g., time spent watching television; LaBrie et al., 2013).
  Interventions: Behavioral: Inhibitory Control Training
- Working Memory Training without Normative Feedback (Experimental): A battery of working memory tasks will be used during the intervention period. These tasks were selected from previous research evaluating working memory training in substance use disorder (Bickel et al., 2011b; Houben et al., 2011b). Tasks will include visuospatial working memory task, digit span task, letter span task, and the n-back task. Subjects assigned to not receive normative feedback will receive feedback on time spent doing a non-alcohol related activity as an attention/informational control (e.g., time spent watching television; LaBrie et al., 2013).
  Interventions: Behavioral: Working Memory Training

INTERVENTIONS:
Behavioral: Normative Feedback — Subjects assigned to normative feedback will be directed to a statement standardized based on subjects' reported average number of standard drinks per week, age, and gender.
  Arms: Attentional Control with Normative Feedback; Inhibitory Control Training with Normative Feedback; Working Memory Training with Normative Feedback
Behavioral: Inhibitory Control Training — The inhibitory control training task is a modified version of the Cued Go/No-Go tasks (Weafer and Fillmore, 2012; Miller et al. 1991) and is based on a task currently used in our laboratory targeting cocaine inhibitory control.
  Arms: Inhibitory Control Training with Normative Feedback; Inhibitory Control Training without Normative Feedback
Behavioral: Working Memory Training — A battery of working memory tasks will be used during the intervention period. These tasks were selected from previous research evaluating working memory training in substance use disorder (Bickel et al., 2011b; Houben et al., 2011b). Tasks will include visuospatial working memory task, digit span task, letter span task, and the n-back task.
  Arms: Working Memory Training with Normative Feedback; Working Memory Training without Normative Feedback

SUMMARY:
The purpose of this study is to test the feasibility and acceptability of delivering cognitive training over mTurk. Subjects will be randomized to a 1) inhibitory control training condition, 2) working memory training condition, or 3) control training condition. Recent studies have also demonstrated the feasibility and potential efficacy of delivering brief normative feedback to reduce alcohol consumption through mTurk. In these brief interventions, subjects are provided information about their drinking compared to their same age and gendered peers. Approximately half of the subjects in each cognitive training group will receive normative feedback to evaluate effects on alcohol consumption and possible interactions with cognitive training. This study will focus on alcohol use given the ease and clinical acceptance of alcohol use self-report as a primary outcome.

DETAILED DESCRIPTION:
Alcohol use disorder is a persistent public health concern. Approximately 16 million Americans met criteria for alcohol use disorder in 2015, with the annual economic impact of excessive drinking estimated at $250 billion. Alcohol use can also interact with other licit (e.g., cigarettes) and illicit (e.g., cocaine) substances to increase health risks . At least half of all violent crimes involve alcohol consumption and problem drinking plays an important role in domestic abuse and intimate partner violence . These evident economic, health, and social implications of alcohol misuse highlight the importance of understanding determinants of alcohol use behaviors and developing interventions designed to address maladaptive patterns of use.

Cognitive training to address alcohol and other substance use disorders has received a great deal of attention in the interventions development literature. Training may be broadly divided into two classes: 1) cognitive bias modification and response inhibition (i.e., inhibitory control) and 2) working memory interventions. Inhibitory control training attempts to retrain prepotent responses away from drug-related cues by specifically pairing those cues with no-go signals in training tasks. Working memory training uses cognitive-behavioral tasks (e.g., letter/digit strings, visual search, n-back) to improve information maintenance and manipulation. These brief interventions hold particular appeal because they may be easily incorporated into comprehensive approaches to substance use treatment. For example, cognitive improvements due to brief training may improve engagement with and attention to cognitive-behavioral therapy and compliance with homework and other program-related activities. Generally speaking, training has consistently demonstrated improvements on the trained or similar tasks as well as related concepts (e.g., delay discounting is improved after working memory training). Improvements in dissimilar tasks or different domains are not consistently observed, however, and clinical measures, such as drug use, have seen mixed outcomes.

A significant limitation of the extant literature is the relatively small samples typically evaluated (i.e., 20-40 subjects per condition). It is likely that the effects of cognitive training are of a small-to-medium effect size, however, the relatively low costs of training procedures mean that small effect sizes may not preclude clinical utility. It is also likely that individual characteristics will moderate the utility of these interventions for impacting substance use or related negative health behaviors. The use of small samples precludes testing these types of moderators with adequate statistical power as does the recruitment of comparably homogeneous samples (e.g., student samples, individuals from a single addiction clinic).

An emerging method addressing these concerns is crowdsourcing. Crowdsourcing, such as on Amazon.com's Mechanical Turk (mTurk), allows for the effective and efficient sampling of diverse subjects. We have previously demonstrated a close correspondence between in-person and online findings using mTurk in substance use research providing support for the validity of the resource. We have also recently demonstrated feasibility, acceptability, and validity of conducting intensive longitudinal research related to substance use on this platform. Demonstrating the feasibility and acceptability of applying cognitive training methods through mTurk would help establish this setting for future large sample studies testing novel interventions and/or individual characteristic moderating intervention efficacy.

The purpose of this study is to test the feasibility and acceptability of delivering cognitive training over mTurk. Subjects will be randomized to a 1) inhibitory control training condition, 2) working memory training condition, or 3) control training condition. Recent studies have also demonstrated the feasibility and potential efficacy of delivering brief normative feedback to reduce alcohol consumption through mTurk. In these brief interventions, subjects are provided information about their drinking compared to their same age and gendered peers. Approximately half of the subjects in each cognitive training group will receive normative feedback to evaluate effects on alcohol consumption and possible interactions with cognitive training. This study will focus on alcohol use given the ease and clinical acceptance of alcohol use self-report as a primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported past week alcohol use.
* Meet criteria for Alcohol Use Disorder (AUD), verified by computerized questionnaire for DSM-V AUD criteria (Appendix A).
* Age 21 years or older.
* Express interest in completing a 2-week study involving daily cognitive tasks.
* Residence in the United States

Exclusion Criteria:

* N/A

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig R Rush, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strickland JC, Hill JC, Stoops WW, Rush CR. Feasibility, Acceptability, and Initial Efficacy of Delivering Alcohol Use Cognitive Interventions via Crowdsourcing. Alcohol Clin Exp Res. 2019 May;43(5):888-899. doi: 10.1111/acer.13987. Epub 2019 Mar 19. PMID 30888705

RESULTS

PARTICIPANT FLOW:
Groups:
- Attentional Control With Normative Feedback: Control training tasks included completion of basic arithmetic problems for approximately 5 minutes. Subjects assigned to normative feedback were directed to a statement standardized based on subjects' reported average number of standard drinks per week, age, and gender.
  Normative Feedback: Subjects assigned to normative feedback will be directed to a statement standardized based on subjects' reported average number of standard drinks per week, age, and gender.
- Inhibitory Control Training With Normative Feedback: The inhibitory control training task is a modified version of the Cued Go/No-Go tasks (Weafer and Fillmore, 2012; Miller et al. 1991) and is based on a task currently used in our laboratory targeting cocaine inhibitory control. Subjects assigned to normative feedback were directed to a statement standardized based on subjects' reported average number of standard drinks per week, age, and gender.
  Normative Feedback: Subjects assigned to normative feedback will be directed to a statement standardized based on subjects' reported average number of standard drinks per week, age, and gender.
  Inhibitory Control Training: The inhibitory control training task is a modified version of the Cued Go/No-Go tasks (Weafer and Fillmore, 2012; Miller et al. 1991) and is based on a task currently used in our laboratory targeting cocaine inhibitory control.
- Working Memory Training With Normative Feedback: A battery of working memory tasks was used during the intervention period. These tasks were selected from previous research evaluating working memory training in substance use disorder (Bickel et al., 2011b; Houben et al., 2011b). Tasks included visuospatial working memory task, digit span task, letter span task, and the n-back task. Subjects assigned to normative feedback were directed to a statement standardized based on subjects' reported average number of standard drinks per week, age, and gender.
- Attentional Control Without Normative Feedback: Control training tasks included completion of basic arithmetic problems for approximately 5 minutes. Subjects assigned to not receive normative feedback received feedback on time spent doing a non-alcohol related activity as an attention/informational control (e.g., time spent watching television; LaBrie et al., 2013).
- Inhibitory Control Training Without Normative Feedback: The inhibitory control training task is a modified version of the Cued Go/No-Go tasks (Weafer and Fillmore, 2012; Miller et al. 1991) and is based on a task currently used in our laboratory targeting cocaine inhibitory control. Subjects assigned to not receive normative feedback received feedback on time spent doing a non-alcohol related activity as an attention/informational control (e.g., time spent watching television; LaBrie et al., 2013).
  Inhibitory Control Training: The inhibitory control training task is a modified version of the Cued Go/No-Go tasks (Weafer and Fillmore, 2012; Miller et al. 1991) and is based on a task currently used in our laboratory targeting cocaine inhibitory control.
- Working Memory Training Without Normative Feedback: A battery of working memory tasks was used during the intervention period. These tasks were selected from previous research evaluating working memory training in substance use disorder (Bickel et al., 2011b; Houben et al., 2011b). Tasks included visuospatial working memory task, digit span task, letter span task, and the n-back task. Subjects assigned to not receive normative feedback received feedback on time spent doing a non-alcohol related activity as an attention/informational control (e.g., time spent watching television; LaBrie et al., 2013).
  Working Memory Training: A battery of working memory tasks will be used during the intervention period. These tasks were selected from previous research evaluating working memory training in substance use disorder (Bickel et al., 2011b; Houben et al., 2011b). Tasks will include visuospatial working memory task, digit span task, letter span task, and the n-back task.
Period: Overall Study
Arm/Group | Attentional Control With Normative Feedback | Inhibitory Control Training With Normative Feedback | Working Memory Training With Normative Feedback | Attentional Control Without Normative Feedback | Inhibitory Control Training Without Normative Feedback | Working Memory Training Without Normative Feedback
Started | 76 | 72 | 76 | 73 | 73 | 74
Completed | 68 | 68 | 66 | 64 | 70 | 66
Not Completed | 8 | 4 | 10 | 9 | 3 | 8
Not completed — Lost to Follow-up | 8 | 4 | 10 | 9 | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Attentional Control With Normative Feedback | Inhibitory Control Training With Normative Feedback | Working Memory Training With Normative Feedback | Attentional Control Without Normative Feedback | Inhibitory Control Training Without Normative Feedback | Working Memory Training Without Normative Feedback | Total
Number analyzed (Participants) | 76 | 72 | 76 | 73 | 73 | 74 | 444
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (8.7) | 32.5 (9.3) | 35.2 (9.5) | 35.8 (11.0) | 34.3 (10.9) | 33.7 (8.5) | 34.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 40 | 41 | 41 | 36 | 30 | 227
  Male | 37 | 32 | 35 | 32 | 37 | 44 | 217
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 6 | 6 | 5 | 1 | 3 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 6 | 4 | 5 | 5 | 28
  White | 62 | 59 | 62 | 61 | 66 | 64 | 374
  More than one race | 3 | 4 | 0 | 3 | 0 | 2 | 12
  Unknown or Not Reported | 1 | 0 | 2 | 0 | 1 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 76 | 72 | 76 | 73 | 73 | 74 | 444

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Use
Description: Self-report of percent of heavy alcohol drinking days
Time Frame: Past two weeks
Population: These data include only participants that were randomized and completed the follow-up assessment providing valid alcohol use data.
Measure: Mean (Standard Deviation); unit: percentage heavy drinking days
Arm/Group | Attentional Control With Normative Feedback | Inhibitory Control Training With Normative Feedback | Working Memory Training With Normative Feedback | Attentional Control Without Normative Feedback | Inhibitory Control Training Without Normative Feedback | Working Memory Training Without Normative Feedback
Number analyzed (Participants) | 50 | 50 | 50 | 51 | 58 | 50
percentage heavy drinking days | 19.4 (30.3) | 16.3 (29.4) | 15.3 (25.0) | 19.1 (29.7) | 19.6 (26.7) | 21.0 (30.7)

2. Secondary Outcome: Percentage of Sessions Completed (Feasibility)
Description: Completion rates during intervention period
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: percentage of sessions completed
Arm/Group | Attentional Control With Normative Feedback | Inhibitory Control Training With Normative Feedback | Working Memory Training With Normative Feedback | Attentional Control Without Normative Feedback | Inhibitory Control Training Without Normative Feedback | Working Memory Training Without Normative Feedback
Number analyzed (Participants) | 76 | 72 | 76 | 73 | 73 | 74
percentage of sessions completed | 68.6 (35.1) | 63.3 (35.5) | 56.5 (39) | 66.1 (35.3) | 74.7 (32.6) | 59.9 (37)

3. Secondary Outcome: Treatment Acceptability Questionnaire
Description: Total average ratings on a treatment acceptability questionnaire, rated from 0 (minimum) to 100 (maximum). Higher scores indicate greater treatment acceptability.
Time Frame: 2 weeks
Population: These data include only participants that were randomized and completed the follow-up assessment providing valid acceptability data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attentional Control With Normative Feedback | Inhibitory Control Training With Normative Feedback | Working Memory Training With Normative Feedback | Attentional Control Without Normative Feedback | Inhibitory Control Training Without Normative Feedback | Working Memory Training Without Normative Feedback
Number analyzed (Participants) | 58 | 58 | 57 | 57 | 64 | 58
units on a scale | 80.8 (18.3) | 75.9 (21.4) | 77.9 (20.9) | 84.2 (19.3) | 81.9 (17.3) | 74.6 (19)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 4 week study period (2 week intervention and 2 week follow-up)
Groups:
- Working Memory Training With Normative Feedback: A battery of working memory tasks was used during the intervention period. These tasks were selected from previous research evaluating working memory training in substance use disorder (Bickel et al., 2011b; Houben et al., 2011b). Tasks included visuospatial working memory task, digit span task, letter span task, and the nback task. Subjects assigned to normative feedback were directed to a statement standardized based on subjects' reported average number of standard drinks per week, age, and gender
- Attentional Control Without Normative Feedback: Control training tasks included completion of basic arithmetic problems for approximately 5 minutes. Subjects assigned to not receive normative feedback received feedback on time spent doing a nonalcohol related activity as an attention/informational control (e.g., time spent watching television; LaBrie et al., 2013).
- Inhibitory Control Training Without Normative Feedback: The inhibitory control training task is a modified version of the Cued Go/No-Go tasks (Weafer and Fillmore, 2012; Miller et al. 1991) and is based on a task currently used in our laboratory targeting cocaine inhibitory control. Subjects assigned to not receive normative feedback received feedback on time spent doing a nonalcohol related activity as an attention/informational control (e.g., time spent watching television; LaBrie et al., 2013). Inhibitory Control Training: The inhibitory control training task is a modified version of the Cued Go/No-Go tasks (Weafer and Fillmore, 2012; Miller et al. 1991) and is based on a task currently used in our laboratory targeting cocaine inhibitory control.
- Working Memory Training Without Normative Feedback: A battery of working memory tasks was used during the intervention period. These tasks were selected from previous research evaluating working memory training in substance use disorder (Bickel et al., 2011b; Houben et al., 2011b). Tasks included visuospatial working memory task, digit span task, letter span task, and the nback task. Subjects assigned to not receive normative feedback received feedback on time spent doing a nonalcohol related activity as an attention/informational control (e.g., time spent watching television; LaBrie et al., 2013). Working Memory Training: A battery of working memory tasks will be used during the intervention period. These tasks were selected from previous research evaluating working memory training in substance use disorder (Bickel et al., 2011b; Houben et al., 2011b). Tasks will include visuospatial working memory task, digit span task, letter span task, and the nback task.
Arm/Group | Attentional Control With Normative Feedback | Inhibitory Control Training With Normative Feedback | Working Memory Training With Normative Feedback | Attentional Control Without Normative Feedback | Inhibitory Control Training Without Normative Feedback | Working Memory Training Without Normative Feedback
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/72 | 0/76 | 0/73 | 0/73 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/72 | 0/76 | 0/73 | 0/73 | 0/74
Other Adverse Events (participants affected / at risk) | 0/76 | 0/72 | 0/76 | 0/73 | 0/73 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT03438539/Prot_SAP_000.pdf